CLINICAL TRIAL: NCT00235365
Title: Metacognitive Therapy for Patients With a Psychiatric Disorder and Comorbid Insomnia.
Brief Title: Metacognitive Therapy for Comorbid Insomnia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: problems recruiting patients
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2005.2.gr
Record Dates: First submitted 2005-10-07; First posted 2005-10-10 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Secondary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- meta-cognitive therapy (Experimental): meta-cognitive therapy
  Interventions: Behavioral: meta-cognitive therapy
- waiting list (Active Comparator): waiting list control
  Interventions: Other: waiting list

INTERVENTIONS:
Behavioral: meta-cognitive therapy — Meta-cognitive therapy
  Arms: meta-cognitive therapy
Other: waiting list — waiting list control
  Arms: waiting list

SUMMARY:
The purpose of this study is to determine the effect of meta-cognitive therapy for insomnia.

DETAILED DESCRIPTION:
This study is a randomized controlled trial with 50 patients with a psychiatric disorder and insomnia. The patients will be randomized into two groups of 25 patients. The first group receives meta-cognitive therapy, whereas the second group will be assigned to a waiting list control.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia secondary to a primary psychiatric disorder

Exclusion Criteria:

* substance abuse, psychotic symptoms, suicidal intentions, severe organic disorder or psychiatric disorder where sleep restriction is not advised, organic sleep disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Scores on rating scales for sleep quality | one year

SECONDARY OUTCOMES:
Scores on rating scales for depression, psychiatric symptom severity, and cognitive processing. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Morken, PhD MD, Principal Investigator — Norwegian University of Science and Technology